CLINICAL TRIAL: NCT00938353
Title: Multicentre, Randomized, Double-blind, Placebo-controlled, Two-arm Parallel Groups Study Design to Demonstrate the Efficacy and Tolerability of a Single Dose of BDP Suspension for Nebulisation 1600 µg vs Placebo in the Treatment of Children Aged 6 Months to 3 Years With a Clinical Diagnosis of Moderate Croup
Brief Title: Efficacy of Nebulized Beclomethasone Dipropionate (BDP) in the Treatment of Moderate Croup
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: possibility to discriminate the active drug from placebo
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Dr. Gabriele Nicolini, Chiesi Farmaceutici S.p.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC/PR/1404/003/09; EUDRACT No. 2009-014376-22
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Croup
Keywords: Moderate croup (Westley score 3-8)
MeSH Terms: conditions — Croup

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BDP UDV (Experimental)
  Interventions: Drug: beclomethasone dipropionate suspension for nebulisation 800 mcg/2 ml
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo solution for nebulisation 2 ml

INTERVENTIONS:
Drug: beclomethasone dipropionate suspension for nebulisation 800 mcg/2 ml — Single dose 1600 mcg/4 ml
  Arms: BDP UDV
Drug: Placebo solution for nebulisation 2 ml — single dose: 4 ml
  Arms: Placebo

SUMMARY:
Acute laryngotracheobronchitis, better known as croup, is one of the common respiratory complaints among children and the most common cause of airway obstruction in children aged six months to six years. Patients with croup are typically visited by physicians during two peak time periods throughout the year. The first one is in the autumn, usually as a result of parainfluenza virus, and the second peak occurs in early winter, a consequence of RSV. Croup affects males more commonly than females and affects children between the ages of 6 months to 6 years. The incidence of croup peaks in children at 2 years of age; croup in older children is uncommon, and recurrent episodes are frequently observed.

Croup symptoms are generally short-lived, with about 60% of children showing resolution of their barky cough within 48 h. However, a few children continue to have symptoms for up to 1 week. Although most children with croup recover without specific treatment, up to 15% require hospital admission, and, among those admitted, up to 5% may require intubation.

Nebulised adrenaline is effective but it has a short duration of action and potentially dangerous side effects, and it is therefore not recommended for use in the community in mild-moderate Croup.

Oral and intramuscular steroid treatment, when given in adequate doses in hospital, has been shown to be effective for moderate to severe croup in a number of trials and a meta analysis.

It has been suggested that nebulised administration is superior to the oral or intramuscular route of administration for a more rapid onset of action and fewer side-effects.

This study is aimed to demonstrate the effectiveness of nebulised steroid administration as beclomethasone dipropionate in croup patients compare to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained by parents/legal representative prior to any study-related procedures.
2. Male or female subject aged between 6 months and 3 years referring to ER with acute onset barky cough, stridor, hoarseness, and respiratory distress
3. Children with a diagnosis of moderate croup (Westley score 3-8)

Exclusion Criteria:

1. Symptoms or signs of any other cause of stridor;
2. Previous acute angioneurotic oedema;
3. Children with diagnosis of severe croup (Wesley score >8);
4. History of congenital or acquired stridor, diagnosis of epiglottitis, chronic pulmonary disease, asthma, severe systemic disease, exposure to chickenpox virus within the previous 21 days, or known immune dysfunction;
5. Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study;
6. Treatment with oral or parenteral corticosteroids within the previous 2 weeks; Treatment with epinephrine for respiratory distress before enrollment;
7. Previous visit to an emergency room department due to croup during this episode of the disease;
8. Inability of the parent to understand the nature and scope of the study or the possible benefits or unwanted effects of the study treatments;
9. Enrollment in another clinical trial in the previous 4 weeks or subject already admitted in this study
10. Lack of a telephone at home;

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate superiority of nebulized BDP vs placebo in Westley croup score at 6 h | 6 h

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Giuseppe Moscati, Avellino, Italy